CLINICAL TRIAL: NCT05386888
Title: A Phase 2 Trial of GFH018 and Toripalimab in Combination With Concurrent Chemoradiotherapy for Patients With Unresectable, Locally Advanced Stage III Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Trial of GFH018 and Toripalimab in Combination With Concurrent Chemoradiotherapy in Stage III NSCLC Chemoradiotherapy in Stage III NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH018X1202
Record Dates: First submitted 2022-05-12; First posted 2022-05-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: NSCLC, Stage III
Keywords: Locally Advanced; Unresectable NSCLC; TGF-βRI; PD-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab; Paclitaxel; Carboplatin; Cisplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Primary Purpose: ORR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): GFH018 80mg 7-Day on/ 7-Day off and 4 doses of Toripalimab 240mg Q3W concurrently with standard chemo-radiotherapy, followed by GFH018 80mg 14-Day on/ 14-Day off and Toripalimab 3mg/kg Q2W for up to 48 weeks
  Interventions: Drug: GFH018; Drug: Toripalimab; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Radiation: Thoracic Radiation Therapy (TRT)

INTERVENTIONS:
Drug: GFH018 — Administered as oral
Drug: Toripalimab — Administered as an IV infusion
Drug: Paclitaxel — Administered as an IV infusion
Drug: Carboplatin — Administered as an IV infusion
Drug: Cisplatin — Administered as an IV infusion
Drug: Pemetrexed — Administered as an IV infusion
Radiation: Thoracic Radiation Therapy (TRT) — Thoracic Radiation Therapy (TRT)
Drug: GFH018 — Administered as an IV infusion

SUMMARY:
This is a phase II trial assessing the efficacy and safety of GFH018 and Toripalimab in combination with concurrent chemoradiotherapy (cCRT) in patients with unresectable, locally advanced, Stage III non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Newly diagnosed, pathologically (histologically or cytologically) confirmed, locally advanced, unresectable stage III NSCLC
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Measurable disease (according to RECIST v1.1 criteria)
* Life expectancy > 6 months

Exclusion Criteria:

* Has small cell lung cancer (SCLC) or tumors with the presence of small cell elements.
* Has received prior treatment (chemotherapy, targeted therapy, or radiotherapy) for Stage III NSCLC
* Prior exposure to immune-mediated therapy, including but not limited to, TGFβ inhibitors, anti CTLA-4, anti-PD-1, anti-PD-L1, and anti PD L2 antibodies.
* Known allergy or hypersensitivity to any of the IPs or any of the IP excipients.
* Patients whose radiation treatment plans are likely to encompass a volume of whole lung receiving ≥20 Gy in total (V20) of more than 35% of lung volume.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From the date of enrolment of the first patient up to 28 months , which is also16 months after the enrolment of the last patient
  Objective response rate (ORR) is defined as the percentage of patients with objective response (OR).
  OR was determined using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). OR is defined as the best overall response (Complete Response (disappearance of all target and non-target lesions; no new lesions) or Partial Response (≥decrease in the sum of the largest diameters of target lesions; no new lesions)) across all assessment points from enrollment to termination of trial treatment. Radiological tumour assessment was performed using CT scans.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No